CLINICAL TRIAL: NCT03817320
Title: A TACL Phase 1/2 Study of PO Ixazomib in Combination With Chemotherapy for Childhood Relapsed or Refractory Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma IND# 140730
Brief Title: PO Ixazomib in Combination With Chemotherapy for Childhood Relapsed or Refractory Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Takeda (Industry); Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2017-002
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: ALL, Childhood; Lymphoblastic Lymphoma, Childhood; Lymphoblastic Leukemia, Acute, Childhood
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ixazomib; Vincristine; Dexamethasone; Asparaginase; Doxorubicin; Methotrexate; Hydrocortisone; Cytarabine; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ixazomib Dose Level 1 (Stratum A) (Experimental): Patients will be treated on ixazomib at 1.6 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15, Doxorubicin at 60 mg/m^2 on Days 1, Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14, and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
  Interventions: Drug: Ixazomib; Drug: Vincristine; Drug: Dexamethasone; Drug: Asparaginase; Drug: Doxorubicin; Drug: Methotrexate (IT); Drug: Triple IT (Methotrexate, Hydrocortisone, Cytarabine)
- Ixazomib Dose Level 2 (Stratum A) (Experimental): Patients will be treated on ixazomib at 2.0 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15, Doxorubicin at 60 mg/m^2 on Days 1, Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14, and IT chemotherapy dependent on patient's CNS status at time of enrollment. Patients will be treated at this arm Dose Level once patient accrual at Dose Level 1 has been completed and dose escalation is allowed as defined by the 3+3 design.
  Interventions: Drug: Ixazomib; Drug: Vincristine; Drug: Dexamethasone; Drug: Asparaginase; Drug: Doxorubicin; Drug: Methotrexate (IT); Drug: Triple IT (Methotrexate, Hydrocortisone, Cytarabine)
- Ixazomib Dose Level -1 (Stratum A) (Experimental): Patients will be treated on ixazomib at 1.2 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15, Doxorubicin at 60 mg/m^2 on Days 1, Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14, and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm Dose Level -1 is needed only if de-escalation from Dose Level 1 is required.
  Interventions: Drug: Ixazomib; Drug: Vincristine; Drug: Dexamethasone; Drug: Asparaginase; Drug: Doxorubicin; Drug: Methotrexate (IT); Drug: Triple IT (Methotrexate, Hydrocortisone, Cytarabine)
- Ixazomib Dose Level 1 (Stratum B) (Experimental): Patients will be treated on ixazomib at 1.6 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15, Doxorubicin at 60 mg/m^2 on Days 1, Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14, and IT chemotherapy dependent on patient's CNS status at time of enrollment. Leucovorin PO/IV at 5 mg/m^2/dose X 2 doses given 24 and 30 hours after IT Methotrexate or Triple IT will also be given on this arm. This arm is only for patients with Down syndrome (Stratum B).
  Interventions: Drug: Ixazomib; Drug: Vincristine; Drug: Dexamethasone; Drug: Asparaginase; Drug: Doxorubicin; Drug: Methotrexate (IT); Drug: Triple IT (Methotrexate, Hydrocortisone, Cytarabine); Drug: Leucovorin

INTERVENTIONS:
Drug: Ixazomib — Days 1, 4, 8, and 11. Note: at least 72 hours must have elapsed between doses
  Dose Phase 1 - Assigned upon study entry.
  Phase 2 - PO formulation at RP2D
Drug: Vincristine — IV push over 1 minute or infusion via minibag as per institutional policy
  Days 1, 8, 15 and 22
  Dose: ≥ 1 year: 1.5mg/m2/dose (maximum dose 2mg)
  ≥ 6 months and < 1 year: 1.2mg/m2/dose
  < 6 months: 1mg/m2/dose
Drug: Dexamethasone — Days 1-14
  Dose: ≥ 1 year: 10mg/m2/day, divided BID (i.e., 5mg/m2/dose, BID)
  ≥ 6 months and < 1 year: 8mg/m2/day, divided BID (i.e., 4 mg/m2/dose, BID)
  < 6 months: 7mg/m2/day, divided BID (i.e., 3.5 mg/m2/dose, BID)
Drug: Asparaginase — Days 2, 15
  Dose ≥ 1 year: 2,500 International units (IU)/m2/dose
  ≥ 6 months and < 1 year: 2,000 IU/m2/dose
  < 6 months: 1,750 IU/m2/dose
  Patient with allergic reaction to Pegaspargase can be given Erwinase IM/IV on Mon/Wed/Fri (or every other day per institutional standard) x 6 doses for each dose of Pegaspargase.
  Dosing guideline for Erwinase:
  * 1 year: 25,000 IU/m2/dose
  * 6 months and < 1 year: 20,000 IU/m2/dose
  < 6 months: 17,500 IU/m2/dose
Drug: Doxorubicin — Day 1
  Dose ≥ 1 year: 60mg/m2/dose
  ≥ 6 months and < 1 year: 48 mg/m2/dose
  < 6 months: 42mg/m2/dose
Drug: Methotrexate (IT) — For patients with CNS 1 or CNS 2, on Days 1, 15, and 29
Drug: Triple IT (Methotrexate, Hydrocortisone, Cytarabine) — For patients with CNS 3, on Days 1, 8, 15, 22, and 29
Drug: Leucovorin — For patients with Down syndrome only, on Days 2, 9, 16, 23, and 30 (based on dates when IT Methotrexate or Triple IT is given)
  Arms: Ixazomib Dose Level 1 (Stratum B)

SUMMARY:
This is a phase 1/2 study of a drug called Ixazomib in combination with cytotoxic chemotherapy consisting of Vincristine, Dexamethasone, Asparaginase, and Doxorubicin (VXLD).

DETAILED DESCRIPTION:
The phase 1 study is to determine the maximum tolerated dose (MTD) of the PO formulation, followed by a screening phase 2 study to investigate the efficacy of ixazomib in combination with chemotherapy in children with relapsed ALL and lymphoblastic lymphoma (LLy). The single arm, screening phase 2 design will allow us to use a minimal number of patients to obtain preliminary information about treatment efficacy. Discovering a safe and tolerable dose of ixazomib in a PO formulation and the preliminary efficacy data will significantly increase the possibility of ixazomib moving forward in frontline pediatric treatment protocols in both intense chemotherapy courses and maintenance courses.

ELIGIBILITY:
Inclusion Criteria:

* Age Patients must be ≤21 years of age at the time of enrollment.

  1. Phase 1 - Initial enrollment will be restricted to patients < 18 years of age until 9 such patients are enrolled
  2. Phase 2 - Initial enrollment will be restricted to patients < 18 years of age until 6 such patients are enrolled (applies to Stratum A only)
* Diagnosis Patients must have a diagnosis of relapsed/refractory ALL or LLy with or without extramedullary disease (including CNS2 and CNS3). Patient with mixed phenotype ALL or mature B (Burkitt-like) leukemia are not eligible.

  1. Patients with ALL must have ≥ 5% blasts by morphology.
  2. Patients with LLy must have measurable disease documented by clinical, radiologic or histologic criteria
* Performance Level Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50% for patients ≤ 16 years of age.
* Prior Therapy A. Prior therapeutic attempts

  * Phase 1 - Any patients with relapsed/refractory ALL or LLy
  * Phase 2

    1. B-cell ALL/LLy: all patients must have failed two or more therapeutic attempts.
    2. T-cell ALL/LLy: all patients must have failed one or more therapeutic attempts. B. Recent prior chemotherapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
  * Myelosuppressive chemotherapy: At least 14 days must have elapsed since the completion of myelosuppressive therapy. However, patients may receive any of the following medications within 14 days without a "wash-out" period:
* Hydroxyurea: Hydroxyurea can be initiated and/or continued for up to 24 hours prior to the start of protocol therapy.

  * "Maintenance-style" therapy - Therapy including vincristine (dosed at a maximum of one-time weekly), oral 6-mercaptopurine, oral methotrexate (dosed at a maximum of one-time weekly), dexamethasone (dosed at ≤ 3 mg*/m^2/dose twice daily), and prednisone (dosed at ≤ 20 mg*/m^2/dose twice daily) can be initiated and/or continued for up to 24 hours prior to the start of protocol therapy.

    * Doses can be rounded to adjust for pill size

C. Hematopoietic stem cell transplant: Patients who have experienced their relapse after a HSCT are eligible, provided they have no evidence of acute or chronic Graft-versus-Host Disease (GVHD), are not receiving GVHD prophylaxis or treatment, and are at least 90 days post-transplant at the time of enrollment.

D. Hematopoietic growth factors: It must have been at least 7 days since the completion of therapy with G-CSF or other growth factors at the time of enrollment. It must have been at least 14 days since the completion of therapy with long-acting filgrastim (pegfilgrastim or biosimilar)

E. Biologic (anti-neoplastic agent): At least 7 days since the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair

1. Monoclonal antibodies: At least 3 half-lives of the antibody or 21 days (whichever is shorter) must have elapsed after the last dose of monoclonal antibody. (i.e., blinatumomab half-life = 6 hours, therefore washout is 18 hours; inotuzumab half-life = 37 days therefore washout is 21 days; rituximab half-life = 66 days, therefore washout is 21 days). If steroids are being used to modify immune-related adverse events of antibody therapy, at least 14 days must have elapsed since the last dose of corticosteroid.
2. Immunotherapy: At least 30 days after the completion of any type of immunotherapy, e.g., tumor vaccines, CAR T cells. If steroids are being used to modify immune-related adverse events of immunotherapy, at least 14 days must have elapsed since the last dose of corticosteroid.

F. XRT: Craniospinal XRT is prohibited during protocol therapy. No washout period is necessary for radiation given to any extramedullary site other than CNS; ≥90 days must have elapsed if prior total body irradiation (TBI) or craniospinal XRT.

G. Anthracyclines: Patients must have had a lifetime exposure of <400 mg/m^2 of doxorubicin equivalents of anthracyclines.

H. Proteasome inhibitors: Patients with a prior exposure to proteasome inhibitors (e.g., bortezomib, carfilzomib) are eligible as long as the patient demonstrated at least a partial response to a proteasome inhibitor with chemotherapy combination. This criteria only applies to the Phase 2 portion of the study.

-Renal and hepatic function

Patients must have adequate renal and hepatic functions as indicated by the following laboratory values:

A. Adequate renal function defined as: Patient must have a calculated creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73m^2 OR a normal serum creatinine based on age/gender

B. Adequate Liver Function Defined as: Direct bilirubin ≤ 1.5 x upper limit of normal (ULN) for age or normal (except in the presence of Gilbert's syndrome), AND alanine transaminase (ALT) ≤ 5 x ULN for age. The hepatic requirements are waived for patients with known or suspected liver involvement by leukemia or lymphoma. This must be reviewed by and approved by the study chair or vice chair.

* Adequate Cardiac Function Defined as: Shortening fraction of ≥ 27% by echocardiogram, OR ejection fraction of ≥ 50% by radionuclide angiogram (MUGA).
* Reproductive Function A. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 2 weeks prior to enrollment.

B. Female patients with infants must agree not to breastfeed their infants while on this study.

C. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment.

* Informed Consent Patients and/or their parents or legal guardians must be capable of understanding the investigational nature, potential risks and benefits of the study. All patients and/or their parents or legal guardians must sign a written informed consent. Age appropriate assent will be obtained per institutional guidelines. To allow non-English speaking patients to participate in this study, bilingual health services will be provided in the appropriate language when feasible.
* All institutional, FDA, and OHRP requirements for human studies must be met.

Exclusion Criteria:

Patients will be excluded if they have isolated CNS or testicular disease.

Patients will be excluded if they have ≥ grade 2 peripheral sensory or motor neuropathy (defined by the Modified "Balis" Pediatric Scale of Pediatric Neuropathies) at the time of enrollment.

Patients will be excluded if they have a known allergy or intolerance to any of the drugs used in the study - except for Pegaspargase for which asparaginase Erwinia chrysanthemi (recombinant)-rywn (Rylaze®) or (if available) crisantaspase (Erwinase®), may be substituted for allergy to Pegaspargase

Patients will be excluded if they have a systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The patient needs to be off pressors and have negative blood cultures for 48 hours.

Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.

Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with the protocol treatment or procedures, interfere with consent, study participation, follow up, or interpretation of study results.

Patients with DNA fragility syndromes (such as Fanconi anemia, Bloom syndrome) are excluded.

Patients will be excluded if they have had a lifetime exposure of ≥400 mg/m2 doxorubicin equivalents of anthracyclines (anthracycline equivalence to doxorubicin conversion see appendix iv) .

Concomitant medications Investigational drugs: Patients currently receiving another investigational drug are not eligible.

Anti-GVHD agents post transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post hematopoetic stem cell transplant are not eligible.

CYP3A4 agents: patients who are currently receiving drugs that are strong inducers of CYP3A4 are not eligible.

Patients with Ph+ALL and Ph-like ALL who are currently receiving TKI therapy

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2025-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Terzah Horton, MD, Study Chair — Baylor College of Medicine
Locations (18):
- United States (17):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas, Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital/Baylor University, Houston, Texas
- The Children's Hospital at Westmead, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixazomib Dose Level 1 (Stratum A): Block 1 - Patients will be treated on ixazomib at 1.6 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15 OR Calaspargase IV 2500 IU/m^2 on Day 2. Doxorubicin at 60 mg/m^2 on Days 1. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
  Block 2 - Patients will be treated on ixazomib at 1.6 mg/m^2/day on Days 1, 4, 8, 15, and 18. Vincristine IV at 1.5 mg/m^2 on Day 3. Pegaspargase IV/IM at 2500 IU/m^2 OR Calaspargase IV 2500 IU/m^2 on Day 9. Methotrexate IV 1000 mg/m^2 on Day 8. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 8.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
- Ixazomib Dose Level 2 (Stratum A): Block 1 - Patients will be treated on ixazomib at 2 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15 OR Calaspargase IV 2500 IU/m^2 on Day 2. Doxorubicin at 60 mg/m^2 on Days 1. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
  Block 2 - Patients will be treated on ixazomib at 2 mg/m^2/day on Days 1, 4, 8, 15, and 18. Vincristine IV at 1.5 mg/m^2 on Day 3. Pegaspargase IV/IM at 2500 IU/m^2 OR Calaspargase IV 2500 IU/m^2 on Day 9. Methotrexate IV 1000 mg/m^2 on Day 8. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 8.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
- Ixazomib Dose Level -1 (Stratum A): Block 1 - Patients will be treated on ixazomib at 1.2 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15 OR Calaspargase IV 2500 IU/m^2 on Day 2. Doxorubicin at 60 mg/m^2 on Days 1. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
  Block 2 - Patients will be treated on ixazomib at 1.2 mg/m^2/day on Days 1, 4, 8, 15, and 18. Vincristine IV at 1.5 mg/m^2 on Day 3. Pegaspargase IV/IM at 2500 IU/m^2 OR Calaspargase IV 2500 IU/m^2 on Day 9. Methotrexate IV 1000 mg/m^2 on Day 8. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 8.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
- Ixazomib Dose Level 1 (Stratum B): Block 1 - Patients will be treated on ixazomib at 1.6 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15 OR Calaspargase IV 2500 IU/m^2 on Day 2. Doxorubicin at 60 mg/m^2 on Days 1. Leucovorin IV/PO at 5 mg/m^2 at hour 24 and 30 post-ITs. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
  Block 2 - Patients will be treated on ixazomib at 1.6 mg/m^2/day on Days 1, 4, 8, 15, and 18. Vincristine IV at 1.5 mg/m^2 on Day 3. Pegaspargase IV/IM at 2500 IU/m^2 OR Calaspargase IV 2500 IU/m^2 on Day 9. Methotrexate IV 1000 mg/m^2 on Day 8. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 8.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
Period: Overall Study
Arm/Group | Ixazomib Dose Level 1 (Stratum A) | Ixazomib Dose Level 2 (Stratum A) | Ixazomib Dose Level -1 (Stratum A) | Ixazomib Dose Level 1 (Stratum B)
Started | 3 | 20 | 0 | 1
Completed | 3 | 18 | 0 | 1
Not Completed | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero patients enrolled on Dose Level -1 of Stratum A as the Dose Level 1 and 2 were deemed safe in Phase I of the study. Dose Level 2 was used as the dose expansion for Phase II. Response-evaluable Stratum A patients treated at the PO RP2D in phase 1 will be included in the phase 2 analysis as per Section 10.1.2 of the study protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixazomib Dose Level 1 (Stratum A) | Ixazomib Dose Level 2 (Stratum A) | Ixazomib Dose Level 1 (Stratum B) | Total
Number analyzed (Participants) | 3 | 20 | 1 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 19 | 1 | 23
  Between 18 and 65 years | 0 | 1 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 1 | 12
  Male | 1 | 11 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 13 | 1 | 16
  Not Hispanic or Latino | 0 | 7 | 0 | 7
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 1 | 11 | 1 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Dose Limiting Toxicity (DLT) During Block 1 of Chemotherapy
Description: The incidence of dose limiting toxicity (DLT) will be measured only during block 1
Time Frame: 5 weeks
Population: Patients with Down Syndrome enrolled in Ixazomib Dose Level 1 (Stratum B) are not eligible for inclusion in the primary DLT or response evaluation. Only the first 6 patients enrolled in Dose Level 2 Stratum A were part of the Phase I portion of this study.
Measure: Count of Participants; unit: Participants
Groups:
- Ixazomib Dose Level 2 (Stratum A): Block 1 - Patients will be treated on ixazomib at 2 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15 OR Calaspargase IV 2500 IU/m^2 on Day 2. Doxorubicin at 60 mg/m^2 on Days 1. Leucovorin IV/PO at 5 mg/m^2 at hour 24 and 30 post-ITs. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
  Block 2 - Patients will be treated on ixazomib at 2 mg/m^2/day on Days 1, 4, 8, 15, and 18. Vincristine IV at 1.5 mg/m^2 on Day 3. Pegaspargase IV/IM at 2500 IU/m^2 OR Calaspargase IV 2500 IU/m^2 on Day 9. Methotrexate IV 1000 mg/m^2 on Day 8. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 8.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
Arm/Group | Ixazomib Dose Level 1 (Stratum A) | Ixazomib Dose Level 2 (Stratum A)
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Primary Outcome: Phase 2: Response (CR + CR MRD-, and CR + CR MRD- + CRi) After Block 1 Chemotherapy at the RP2D
Description: The count of participants below represents the number of patients who achieved CR MRD- or CRi MRD- at the end of block 1 treatment and treated at RP2D (recommended phase 2 dose).
Time Frame: End of Block 1 treatment, Day 29-35 of treatment, assessed within 35 days from treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Dose Level 2 (Stratum A)
Number analyzed (Participants) | 18
Participants | 10

ADVERSE EVENTS:
Time Frame: Adverse events and suspected adverse reactions (CTCAE v5.0 grades 1-5) will be collected and reported from first dose of study therapy through 30 days after the last dose (up to approximately 8 weeks per participant)
Description: No patients enrolled on Dose Level -1 Stratum A. Adverse events were monitored from the first dose of study treatment through 30 days after the last dose for each participant. Response-evaluable Stratum A patients treated at the PO RP2D in phase 1 will be included in the phase 2 analysis as per Section 10.1.2 of the study protocol.
Groups:
- Ixazomib Dose Level 1 (Stratum A): Block 1 - Patients will be treated on ixazomib at 1.6 mg/m^2/day on Days 1, 4, 8, and 11. Vincristine IV at 1.5 mg/m^2 on Days 1, 8, 15 and 22. Pegaspargase IV/IM at 2500 IU/m^2 on Days 2 and 15 OR Calaspargase IV 2500 IU/m^2 on Day 2. Doxorubicin at 60 mg/m^2 on Days 1. . Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 14.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
  Block 2 - Patients will be treated on ixazomib at 1.6 mg/m^2/day on Days 1, 4, 8, 15, and 18. Vincristine IV at 1.5 mg/m^2 on Day 3. Pegaspargase IV/IM at 2500 IU/m^2 OR Calaspargase IV 2500 IU/m^2 on Day 9. Methotrexate IV 1000 mg/m^2 on Day 8. Dexamethasone IV/PO at 10 mg/m^2 continuous starting on Day 1 thru Day 8.and IT chemotherapy dependent on patient's CNS status at time of enrollment. This arm is the starting Dose Level for patients being enrolled.
Arm/Group | Ixazomib Dose Level 1 (Stratum A) | Ixazomib Dose Level 2 (Stratum A) | Ixazomib Dose Level 1 (Stratum B)
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/20 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 14/20 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 20/20 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib Dose Level 1 (Stratum A) (N=3) | Ixazomib Dose Level 2 (Stratum A) (N=20) | Ixazomib Dose Level 1 (Stratum B) (N=1)
Abominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 7 | 0
Allergic Reaction (Immune system disorders) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 7 | 0
Bacteremia (Infections and infestations) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0
Edema Cerebral (Nervous system disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 6 | 0
GGT Increased (Investigations) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 7 | 1
Septic shock (Infections and infestations) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Typhlitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib Dose Level 1 (Stratum A) (N=3) | Ixazomib Dose Level 2 (Stratum A) (N=20) | Ixazomib Dose Level 1 (Stratum B) (N=1)
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 6 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 6 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 11 | 0
Alkaline phosphatase increased (Investigations) | 3 | 5 | 1
Allergic reaction (Immune system disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 16 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 7 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 12 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0
Bleeding labial skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 5 | 0
Blood bilirubin increased (Investigations) | 0 | 10 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0
Buttock Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 3 | 0
Cholesterol high (Investigations) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 5 | 0
Mottled Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
CPK increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0
Decreased Respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 7 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Edema face (General disorders) | 0 | 3 | 0
Edema limbs (General disorders) | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0
Enterocolitis infectious (Gastrointestinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
ERYTHEMATOUS FACIAL RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 0
Fever (General disorders) | 1 | 7 | 0
Fibrinogen decreased (Investigations) | 0 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Eye disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Generalized edema (General disorders) | 0 | 1 | 0
Genital edema (Reproductive system and breast disorders) | 0 | 1 | 0
GGT increased (Investigations) | 0 | 4 | 0
Glucosuria (Renal and urinary disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 4 | 0
Hematuria (Renal and urinary disorders) | 0 | 2 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 12 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 5 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 7 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 9 | 0
Hypertension (Cardiac disorders) | 0 | 6 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 13 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 13 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 6 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 9 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 6 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 18 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 12 | 0
Hypotension (Vascular disorders) | 0 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Increased hunger (General disorders) | 0 | 1 | 0
Increased Respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Increased salivation (General disorders) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
INR increased (Investigations) | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Irritability (Psychiatric disorders) | 1 | 2 | 0
Lactate increased (Investigations) | 0 | 1 | 0
Lesion on left thumb (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 3 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 17 | 0
Methemoglobinemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 5 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 11 | 0
Necrotic Bowel (Gastrointestinal disorders) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 15 | 1
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
irritated PAC Site (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Pain (General disorders) | 1 | 2 | 0
Pale (General disorders) | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
PARAINFLUENZA 1 (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
PARVOVIRUS (Infections and infestations) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Periorbital edema (Eye disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2 | 0
PERIRECTAL BREAKDOWN (Gastrointestinal disorders) | 0 | 1 | 0
PITYROSPORUM FOLLICULITIS (FOREHEAD) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 3 | 14 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
POSITIVE MRSA (Infections and infestations) | 0 | 1 | 0
PRESSURE INJURY (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 2 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RHINOVIRUS (Infections and infestations) | 0 | 1 | 0
SCLERAL HEMORRHAGE (Eye disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 6 | 0
Skin infection (Infections and infestations) | 0 | 2 | 0
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
SYNDROME OF INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 1
Thrombus (Vascular disorders) | 0 | 1 | 0
Thrush (Infections and infestations) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vomiting (Metabolism and nutrition disorders) | 2 | 12 | 0
Weight gain (Metabolism and nutrition disorders) | 0 | 1 | 0
Weight loss (Metabolism and nutrition disorders) | 1 | 1 | 0
White blood cell decreased (Investigations) | 3 | 17 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT03817320/Prot_SAP_ICF_000.pdf